CLINICAL TRIAL: NCT05277701
Title: Lazertinib for Patients With NSCLC Harboring Uncommon EGFR Mutations: A Single-arm, Phase II Multi-center Trial
Brief Title: Lazertinib for Patients With NSCLC Harboring Uncommon EGFR Mutations
Acronym: LU21-16
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1595
Record Dates: First submitted 2022-02-25; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: NSCLC
MeSH Terms: interventions — lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lazertinib (Experimental)
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib — Lazertinib 240mg daily (1 cycle of 21 days) will be applied to the all patients until documented evidence of disease progression, unacceptable toxicity, noncompliance, or withdrawal of consent, or the investigator decides to discontinue treatment, whichever comes first. However, beyond disease progression is allowed based on the investigator's decision. Doses should be taken approximately 24 hours apart at the same time point each day before eating meal under fasting. If it is more than 12 hours after the dose time, the missed dose should not be taken, and patients should be instructed to take the next dose at the next scheduled time.

SUMMARY:
The primary objective is to evaluate the antitumor efficacy of lazertinib in patients with NSCLC harboring uncommon EGFR mutations. The primary endpoint is objective response rate (ORR), defined as the proportion of patients achieving a complete response or partial response per RECIST v1.1 by investigator's assessments.Secondary endpoints are disease control rate, progression-free survival, overall survival, and duration of response. Secondary objectives are progression-free survival, overall survival, and safety profile according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

* Progression-free survival :From C1D1 to the date of either disease progression or death
* Overall survival: From C1D1 to the date of all-cause mortality
* Safety: Evaluated by NCI-CTCAE v5.0
* The exploratory objective is to identify the acquired resistance mechanism to lazertinib in NSCLC with uncommon EGFR mutation.

Lazertinib 240mg daily (1 cycle of 21 days) will be applied to the all patients until documented evidence of disease progression, unacceptable toxicity, noncompliance, or withdrawal of consent, or the investigator decides to discontinue treatment, whichever comes first. However, beyond disease progression is allowed based on the investigator's decision. Doses should be taken approximately 24 hours apart at the same time point each day before eating meal under fasting. If it is more than 12 hours after the dose time, the missed dose should not be taken, and patients should be instructed to take the next dose at the next scheduled time.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer which is not amenable to treatment with a curative aim (e.g. surgery or radiation).
2. Confirmed uncommon EGFR mutations (e.g. G719X, S768I, L861Q, G719X + S768I, G719X + L861Q, L861Q + S768I, L747S, S720A, E709A, exon 18 deletion) without common EGFR mutations including exon 19 deletion, L858R, exon 20 insertion, or T790M. (The result from both cell-free DNA or tissue-based DNA is allowed.)
3. Age of 20 or more.
4. Performance status of Eastern Cooperative Oncology Group 0 to 2.
5. At least one measurable lesion by RECIST 1.1(The part of radiation treatment in the palliative setting is excluded.)
6. Untreated asymptomatic brain metastasis or symptomatic brain metastasis treated with local treatment such as operation, whole brain radiotherapy, or gamma-knife surgery, and stable and not requiring steroids for at least 2 weeks prior to start of study treatment.
7. At least 2 weeks later after whole brain radiotherapy or palliative thoracic radiotherapy
8. Adequate organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; hemoglobin > 9.0g/dL; platelets > 100 x 109/L; total bilirubin ≤1.5 UNL; AST and/or ALT < 2.5 ULN if no demonstrable liver metastases or < 5 UNL in the presence of liver metastases; CCr ≥ 50mL/min
9. Written informed consent form

Exclusion Criteria:

1. Previously treatment with any kind of EGFR TKI
2. Uncontrolled central nervous system metastases
3. Leptomeningeal carcinomatosis
4. Uncontrolled systemic illness, including uncontrolled hypertension, active bleeding, or active infection
5. Cytotoxic chemotherapy, investigational agents or other anticancer drugs within 14days of first dose of study treatment, or any investigational drugs within 5 x half-lives of the compound
6. Major surgery undertaken less than 4 weeks before the study
7. Localized palliative radiotherapy unless completed more than 2 weeks before the study
8. Pregnant or nursing women (Women of reproductive potential have to agree to use an effective contraceptive method, contraception until 3 months after discontinuation of drug for female, hormonal methods should be used in combination with barrier methods)
9. Prior history of malignancy within 5 years from study entry except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, well-treated thyroid cancer, early gastric cancer or otherwise confirmed as curative malignancy disease by principal investigator
10. Any of the following cardiac criteria:

    * Prolonged QT interval in ECG (QTc > 450 msec)
    * Any clinically important abnormalities in rhythm, conduction conduction or morphology of resting ECG eg complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec
    * Any other factors that increase risk of QT or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 yers og age in first degree relatives or concomitant medications known to prolong QT interval

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  It is evaluated by taking CT of the chest and abdomen (including liver and adrenal glands) or MRI .

SECONDARY OUTCOMES:
Progression-free survival(PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS is measured from the date of start of study to the date of disease progression or death from any cause.
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  OS is measured from the date of start of study to the date of death from any cause.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Safety and toxicity profile evaluated throughout the study participation period.

CONTACTS AND LOCATIONS:
Overall Officials: MinHee Hong, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea